CLINICAL TRIAL: NCT02207985
Title: Non Myeloablative Allogeneic Stem Cell Transplantation as Adjuvant Treatment in Patients With Pancreatic Adenocarcinoma
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation in Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Competing studies.
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Brigitta Omazic, M.D, PhD, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANCHSCT
Record Dates: First submitted 2014-06-18; First posted 2014-08-04 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; Hematopoietic stem cell transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hematopoetic stem cell transplantation (Experimental): Patients with pancreatic adenocarcinoma that have undergone Whipple surgery and show no sign of disease recurrence can be treated with hematopoietic stem cell transplantation to achieve an immunological anti-tumor effect.
  Interventions: Procedure: Allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Allogeneic hematopoietic stem cell transplantation

SUMMARY:
Aim:

To study the antitumour effect of reduced intensity conditioning (RIC) with allogeneic stem cell transplantation (HSCT) in patients with pancreatic adenocarcinoma after radical resection of the tumour and adjuvant treatment with standard chemotherapy.

Importance:

If investigators can accomplish an anti-tumour effect using RIC with HSCT as adjuvant treatment in patients with pancreatic adenocarcinoma, it might increase the survival or even cure patients in this group with very poor prognosis.

Primary scientific question:

Can investigators demonstrate an anti-tumour effect against pancreatic adenocarcinoma using adjuvant treatment with HSCT?

Can investigators demonstrate an anti-tumour effect against pancreatic adenocarcinoma using adjuvant treatment with HSCT?

DETAILED DESCRIPTION:
Background Cancer of the pancreas is one of the most common cancer forms in Sweden. Nine-hundred persons receive this diagnosis every year. The 5-year survival is very low, between 5 and 15%, even in the cases where radical resection of the tumor can be performed. This is probably due to minimal residual disease that cannot be diagnosed at the time of surgery. It has recently been shown that micrometastases of pancreatic adenocarcinoma can be detected in tissue samples from lymph nodes and bone marrow, using new sensitive immunohistological methods. When radical resection of the tumour is performed, no microscopically visible tumour is left, but even in this situation, local recurrence of the disease is the most common cause of death in these patients. None of the so far studied adjuvant treatments, irradiation or chemotherapy, has substantially improved the survival in patients with pancreatic adenocarcinoma.

Allogeneic hematopoietic stem cell transplantation (HSCT) is an established curative treatment for malignant blood diseases, mainly leukemia. Using the conventional form of HSCT, where the patient undergoes a myeloablative conditioning with chemotherapy and irradiation, will diminish the amount of malignant cells, but also create space in the bone marrow for the donated stem cells. The myeloablative conditioning induces severe toxic effects, but the patient is rescued by the transplantation of the donated hematopoietic stem cells. The new stem cells will mature into an immune system that will react with the patient's cells, an effect called graft-versus-host reaction (GVHD). It has been shown that the graft-versus-host reaction correlates well with the curative anti-tumor effect. A mild GVH reaction will diminish the risk of relapse, while a severe GVH reaction might be mortal. This anti-tumour effect is mediated by white blood cells of the T-cell type. From this knowledge, the HSCT technique has been developed and nowadays it is possible to use reduced intensity conditioning (RIC). With reduced intensity conditioning using milder forms of chemotherapy, the toxic effects can be reduced, but the immunosuppressive effect is enough to make sure that the hematopoietic stem cells will engraft. Using RIC has lead to treatment of older patients and the anti-tumor effect is just as efficient as with the myeloablative conditioning.

Recently, RIC with HSCT has been used as adjuvant treatment against solid tumours, mainly kidney cancer, colon cancer and breast cancer. An important part of the treatment consists of additional infusion of donor lymphocyte infusions (DLI) after the transplantation to maintain or increase the anti-tumour effect. At our clinic, we have treated about 50 patients with solid tumours using RIC with HSCT. Most of our patients had kidney or colon cancer (19 and 16 patients, respectively), but also two patients with prostate cancer have been treated. About ten patients with primary liver cancers have been treated with liver transplantation combined with RIC with HSCT. The transplantation-related mortality in these patients is about 10-15%.

Aim:

To study the antitumour effect of RIC with HSCT in patients with pancreatic adenocarcinoma after radical resection of the tumour and adjuvant treatment with standard chemotherapy.

Importance:

If investigators can accomplish an anti-tumour effect using RIC with HSCT as adjuvant treatment in patients with pancreatic adenocarcinoma, it might increase the survival or even cure patients in this group with very poor prognosis.

Primary scientific question:

Can investigators demonstrate an anti-tumour effect against pancreatic adenocarcinoma using adjuvant treatment with HSCT?

Secondary scientific questions:

What side-effects will the patient suffer? Can survival be improved compared to standard treatment of pancreatic adenocarcinoma? Is it possible to improve the results by using cytotoxic T-cells against specific pancreatic adenocarcinoma antigens? Are there methods to identify the patients that will have the best results from the treatment? How will quality of life be affected?

Study plan:

The aim of the study is to evaluate the anti-tumour effect of treatment with RIC with HSCT in patients with pancreatic adenocarcinoma. All patients will undergo curative surgery with radical resection of the tumour and adjuvant standard chemotherapy with gemcitabine. HSCT will be offered to patients with an HLA-identical sibling, a kind of biological randomisation. The control group will consist of patients without an HLA-identical sibling, or those declining HSCT.

Inclusion criteria:

Patients with radically resected pancreatic adenocarcinoma that have received adjuvant treatment with standard chemotherapy after surgery.

Exclusion criteria:

Pancreatic adenocarcinoma with metastases or non-radical resection of the tumour. Relapse during standard chemotherapy. Age above 70 years. Severe heart conditions, liver disease, impaired kidney function or other organ dysfunction that will result in severe toxic effects of the HSCT treatment.

Group A will undergo radical resection of the tumour and standard chemotherapy. About eight months after surgery, they will undergo conditioning with cyclophosphamide and fludarabine before transplantation of donated hematopoietic stem cells from their HLA-identical sibling donors. The immunosuppressive treatment, which is given to diminish GVHD, will be tapered quickly to make sure that the anti-tumour effect is as efficient and as fast as possible. Further infusion of DLI will be given to increase or maintain anti-tumour effect in the cases where the graft-versus-host reaction is missing or is very mild. The first DLI will be given intravenously and the second one will be given in A. hepatica to induce a better local effect, since metastases to the liver is a very common event. Conditioning and HSCT will be performed at Centre for Allogeneic Hematopoietic Stem Cell Transplantation and that is also where the follow-up of the patients will be performed. The surgical follow-up will be at the surgical department. Group B will be treated with standard chemotherapy according to current protocols at the department of oncology.

The clinical and laboratory parameters that will be registered are:

* Mortality
* Morbidity
* Time to relapse, will be controled with CT scans
* Quality of life
* Tumour markers
* Detection of cytotoxic T-lymphocytes that have the ability to react with pancreactic adenocarcinoma from the patient as well as cell lines in vitro
* Detection of micrometastases in bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic adenocarcinoma who have undergone curative surgery ad modum Whipple with radical resection of the tumor, R0 or R1.

Exclusion Criteria:

* Pancreatic adenocarcinoma with metastasis or non-radical resection.
* Recurrence of the malignancy after curative surgery and adjuvant chemotherapy.
* Age above 70 years.
* Severe heart disease, liver disease, impaired renal function or other organ failure or underlying diseases that would exclude the patient from undergoing hematopoietic stem cell transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
disease free survival | Five years

CONTACTS AND LOCATIONS:
Locations (1):
- Center for allogeneic stem cell transplantation, Karolinska University hospital, Stockholm, Sweden